CLINICAL TRIAL: NCT01672034
Title: Impact of Laparoscopic Gastric Bypass Surgery and Weight Reduction an Lower Esophageal Sphincter. A Study of Morbidly Obese Patients Before and After Surgery.
Brief Title: Impact of Laparoscopic Gastric Bypass Surgery and Weight Reduction on Lower Esophageal Sphincter (LES)
Status: Withdrawn | Type: Observational
Why Stopped: no patient enrolled
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Alex de Leon, PhD, Specialist in Anaesthesia and Intensive Care, Örebro University, Sweden
Other Study IDs: 2011/477
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese, BMI > 35
  Interventions: Procedure: Laparoscopic gastric bypass surgery

INTERVENTIONS:
Procedure: Laparoscopic gastric bypass surgery

SUMMARY:
The purpose with this study is to investigate whether gastric bypass surgery and the following weight reduction impact the tone in esophageal sphincters and the esophageal function.

In a previous study our group used high resolution solid-state manometry to investigate the pressure in the esophagus and esophageal sphincters in obese patients going through laparoscopic bariatric surgery. These studies showed that the barrier pressure between the stomach and esophagus is significantly lower in obese compared to lean patients. In this study the investigators will examine these patients once more, now after weight reduction to see whether the barrier pressure is back to normal compared to lean patients.

DETAILED DESCRIPTION:
The prevalence of obesity has increased dramatically in recent decades. The gastrointestinal changes associated with obesity have clinical significance for the anesthesiologist in the perioperative period. The upper and lower esophageal sphincters (UES and LES) play a central role in preventing regurgitation and aspiration. The barrier pressure, defined as the difference between the LES pressure and the Intragastric pressure is known to be lower in obese patients compared to lean patients. This might result in a higher risk of regurgitation and aspiration of stomach contents in during induction of anesthesia.

Some studies are made on patients before and after bariatric surgery but results are sparse. In this study the investigators will examine 30 patients before and after bariatric surgery. Our group have performed the measurements on patients before surgery and presented the results in another article. Those patients will be asked to take part of another measurement now 12-18 months after surgery.

30 patients will be consecutively asked and enrolled in this study. Measurements will be performed using high-resolution-solid state manometry.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year,
* BMI prior to surgery > 35,
* ASA-classification 1-3

Exclusion Criteria:

* Patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The initial measurements were made on a group of male and female patients 18-60 years with BMI > 35, ASA-classification 1-3 planned for laparoscopic bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Variation in lower esophageal sphincter tone due to bariatric surgery and weight reduction | 12-18 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive care, University Hospital of Örebro, Örebro, Sweden